CLINICAL TRIAL: NCT02971800
Title: Evaluation of Sodium Fluorescein Use During Intraoperative Cystoscopy After Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Dr Philippe Y Laberge, Gynecologist, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUO-HTL
Record Dates: First submitted 2016-11-15; First posted 2016-11-23 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Ureteral Injury
Keywords: sodium fluorescein; ureteral efflux; laparoscopic hysterectomy
MeSH Terms: interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sodium fluorescein (Experimental): Once hysterectomy completed, a 10 % solution of sodium fluorescein at a 0,25 ml dose (25 mg) is injected before performing diagnostic cystoscopy for all patient.
  Name: Fluorescite Injection 10%, contains sodium fluorescein (equivalent to fluorescein 10% w/v) Dosage : 25 mg Frequency: only once
  Interventions: Drug: sodium fluorescein injection 10%

INTERVENTIONS:
Drug: sodium fluorescein injection 10%
  Other Names: Fluorescite; National Drug Code (NDC) 0065-0092-65

SUMMARY:
The primary objective is to describe the safety and efficacy of intravenous sodium fluorescein to visualize ureteral efflux during intraoperative cystoscopy after total laparoscopic hysterectomy. Secondary objective is to report on surgeon's satisfaction with the overall use of sodium fluorescein.

DETAILED DESCRIPTION:
Thirty patients (n=30) ongoing a total laparoscopic hysterectomy in a tertiary gynecological reference center will be included in this prospective descriptive study.Once hysterectomy is completed, a 10 % solution of sodium fluorescein at a 0,25 ml dose will be injected before performing diagnostic cystoscopy. Time from injection to fluorescent visualization will be recorded as well as coloration density. Adverse events are collected in the operating room, in the recovery room, before patient's discharge and through a home survey.

ELIGIBILITY:
Inclusion Criteria:

* total laparoscopic hysterectomy

Exclusion Criteria:

* breastfeeding
* renal insufficiency
* Medication: Probenecid, digoxin, quinidine, beta-blocker
* hypersensitivity or intolerance to sodium fluorescein

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-08; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Y Laberge, doctorate, Principal Investigator — CHU de Quebec
Locations (1):
- CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants signed informed consent
  1 patient excluded - protocol violation (had laparotomy instead of anticipated laparoscopy)
  1 patient - withdrawal by subject before surgery
  1 patient - excluded before surgery (took an unauthorized drug) 4 patients - excluded before surgery (number needed (30) already reached)
Groups:
- Sodium Fluorescein: Once hysterectomy completed, a 10 % solution of sodium fluorescein at a 0,25 ml dose (25 mg) is injected before performing diagnostic cystoscopy for all patient.
  Name: Fluorescite Injection 10%, contains sodium fluorescein (equivalent to fluorescein 10% w/v) Dosage : 25 mg Frequency: only once
  sodium fluorescein injection 10%
Period: Overall Study
Arm/Group | Sodium Fluorescein
Started | 37
Completed | 30
Not Completed | 7
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Exclusion criteria prior intervention | 1
Not completed — Number evaluable participant already reached | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Fluorescein
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 30
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25 (4)
Surgery duration (min) [Mean (Standard Deviation); unit: minutes] | 141 (47)
Uterus Weight (g) [Mean (Standard Deviation); unit: gram] | 320 (218)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Ureteral Efflux Coloration With Sodium Fluorescein Collected With Dedicated Questionnaire
Description: Time of visualisation of turbulence, time of visualisation of coloration and quality of ureteral efflux coloration (clearly visible or somewhat visible or not visible)
Time Frame: within 15 minutes after the beginning of cystoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Fluorescein
Number analyzed (Participants) | 30
Participants
  Bilateral Coloration clearly visible | 23
  Unilateral Coloration clearly visible and unilateral somewhat visible | 4
  Unilateral Coloration clearly visible (unilateral not visible and no turbulence) | 1
  Bilateral Coloration somewhat visible | 1
  Bilateral Coloration not visible (bilateral turbulence) | 1

2. Primary Outcome: Adverse Reaction Related to Sodium Fluorescein Injection
Time Frame: From sodium fluorescein injection to follow-up 2 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Fluorescein
Number analyzed (Participants) | 30
Participants
  Post-administration hypotension requiring medication | 3
  Sustained nausea in recovery room | 1
  Persistant fluorescent urine coloration at 48 hours | 15
  Itching | 3
  Yellowish skin coloration | 1

3. Secondary Outcome: Surgeon Satisfaction Regarding Ureteral Efflux Visualization by Filling Out a Dedicated Questionnaire
Description: For each participant, surgeon had 3 options to evaluate their satisfaction regarding ureteral efflux coloration with sodium fluorescein during the surgery : very satisfied or satisfied or unacceptable
Time Frame: after cystoscopy (up to 15 min after injection)
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Fluorescein
Number analyzed (Participants) | 30
Participants
  Very satisfied | 27
  Satisfied | 2
  Unacceptable | 1

ADVERSE EVENTS:
Arm/Group | Sodium Fluorescein
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Fluorescein (N=30)
Partial ureteral obstruction (Injury, poisoning and procedural complications) | 1 (1) — 1 participant had a partial ureteral obstruction (13 days after surgery) even if a normal ureteral patency was initially diagnosed. However, the gap between the two jets was the longest observed (6 minutes) in our cohort.
Vault hematoma (Surgical and medical procedures) | 1 (1)
partial vaginal cuff dehiscence (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Fluorescein (N=30)
Sustained nausea (General disorders) | 1 (1)
Yellowish skin coloration (Skin and subcutaneous tissue disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Persistant fluorescent urine coloration (Renal and urinary disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No